CLINICAL TRIAL: NCT02208869
Title: Prospective Russian Study Evaluating the Extent of Underdiagnosed and Undertreated of Familial Hypercholesterolaemia in the Population
Brief Title: Russian Familial Hypercholesterolemia Registry
Acronym: RuFH
Status: Recruiting | Type: Observational
Sponsor: Russian Cardiology Research and Production Center (Other)
Collaborators: Pfizer (Industry); Amgen (Industry); AstraZeneca (Industry)
Responsible Party: Principal Investigator, Marat Vladislavovich Ezhov (MV Ezhov, MD, PhD, DMSc), Leading Researcher, MD, DMSc, Russian Cardiology Research and Production Center
Other Study IDs: SSCRES0179
Record Dates: First submitted 2014-08-02; First posted 2014-08-05 (Estimated); Last update posted 2022-11-02 (Actual); Status verified 2022-11

CONDITIONS: Familial Hypercholesterolemia
Keywords: familial hypercholesterolemia; cholesterol; prevention; registry; atherosclerosis; treatment; prevalence
MeSH Terms: conditions — Hyperlipoproteinemia Type II; Atherosclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Biospecimen Retention: Samples With DNA — whole blood, serum, white cells, urine
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Patients diagnosed with FH: Subjects of both sexes above the age of 18 with TC ≥7.5 mmol/L or LDL-C ≥4.9 mmol/L will be included in the Program. Clinical diagnosis of FH will be established using both the Dutch and the British criteria.
  Those with secondary causes of hypercholesterolemia, such as untreated diabetes mellitus (HbA1c >8%) or hypothyroidism (thyroid-stimulating hormone >1.5 upper normal limit), renal failure (creatinine clearance <30 ml/min), holestatic liver diseases, including biliary cirrhosis, tumors with an active process in the last 5 years will be excluded from the study.

SUMMARY:
True prevalence of FH in the Russian Federation is unknown which leads to low percentage of diagnosed and treated cases. Research is needed to determine the prevalence of FH, specific diagnostic algorithms and optimal treatment strategies. The main aim of the present study is to evaluate the extent to which FH is underdiagnosed and undertreated in the Russian Federation for reduction of cardiovascular risk related to atherosclerosis in the country.

As a first step, total cholesterol (TC) and low-density lipoprotein (LDL-C) levels will be determined in a random sample from Moscow population (n=18000). It is expected that TC ≥ 7.5 mmol/L will be detected in 10% of cohort. During 2014, approximately 500 patients will pass through non-invasive clinical examination at the Russian Cardiology Research and Production Center, including patient demographics, past medical history, family history of hypercholesterolemia, physical findings, current lipid-lowering therapies, blood tests, genetic analysis, echocardiography, carotid duplex ultrasound and exercise SPECT imaging in selected cases. On the basis of the Moscow Program four major Federal Medical Centers will be involved, and FH Registry will be created as a national, multi-center initiative to screen FH patients, control their diagnosis and management, and track clinical-reported outcomes over time.

Establishment of National Guidelines for the diagnosis and treatment of FH on the basis of these data and implementation those into clinical practice in different regions of Russia will allow improving patient care. As an expected outcome, this program will raise awareness and increase appropriate assessment and treatment of FH patients in Russia, leading to a timely detection of the disease and therapy initiation.

DETAILED DESCRIPTION:
*Design. We have chosen a randomly selected cohort of individuals who have been tested in the Moscow office of the "INVITRO" Laboratory on the basis of advertising campaign held in September, 2013, for the purpose of TC level measurement and determination of cardiovascular risk with the use of SCORE chart. The operator from the "INVITRO" Laboratory identified potential FH patients based on TC (≥7.5 mmol/L) or LDL-C (≥4.9 mmol/L) values.

Following identification, the potentially eligible participants suspected for FH are sent a notification letter describing the patient's high cholesterol level, at-atherosclerosis risk status and need for additional screening on the basis of the Russian Cardiology Research and Production Center. Those who give preliminary agreement for participation in the Program are invited to the Institution, where, after signing the ICF, they will undergo clinical (biochemical, echo, duplex scan) and genetic testing. Those individuals refusing to participate in the Program will be taken into account with fixing the reason of unwillingness to participate.

Patients under the age of 18 will be enrolled only with the explicit consent of a parent or legal guardian. All participants will be provided with the information about the Russian FH Community and Russian FH Registry.

All included subjects will be provided with a screening questionnaire querying the patient demographics, past medical history, patient FH history and diagnosis with FH type heterozygous or homozygous, family history of hypercholesterolemia, physical examination findings, current lipid-lowering therapies, and patients' contact information for further follow-up. After initialization of online data capture form (Electronic Medical System), the information will be also entered in the system. Blood and gene banks will be formed; analysis of echocardiography data for aortic valve stenosis, carotid duplex ultrasound for atherosclerosis burden, and exercise SPECT imaging in selected cases of suspected coronary heart disease (CHD) will be performed during the baseline visit. Patients diagnosed with FH on the basis of Dutch Lipid Clinic Network, Simon Broome Criteria and genetic testing will be provided information about screening of first-degree relatives, and additional educational materials about FH (under development).

To determine the true number of heterozygous forms among individuals with a probable diagnosis of FH molecular genetic testing is planned. When a causative mutation is found in the index case, a genetic test will be offered to all first-degree relatives.

Enrolled patients will be asked to update information at annually intervals. Since the last date of data entry, occurrence of major adverse cardiovascular events (acute coronary syndromes, stroke, myocardial revascularization, peripheral revascularization, cardiovascular death), changes in medications, hospitalizations to any reasons, genetic testing, laboratory values, and all-cause mortality will be reviewed.

Follow-up data will be collected yearly following initial enrollment. Updated information on quality of life will be collected. Annual reminder emails will be sent to all patients to call the following physician.

We estimate that at one site during one year (2014-2015) we will screen 500 patients eligible for the participation from the potentially eligible 1505 selected from 18000 individuals.

* Five leading Federal Medical Centers in different regions of Russia will be involved at the first two steps of the Program:

  1. Federal State Institution "Russian Cardiology Research and Production Center" of the Health Ministry of the Russian Federation (Moscow); First line Federal Medical Centers
  2. Samara State Medical University (Samara);
  3. Research Institute of Internal Medicine (Novosibirsk);
  4. Saint-Petersburg State University (Sokolov Center for atherosclerosis and lipid disorders in Clinical Hospital №122 (Saint Petersburg));
  5. Chelyabinsk State Medical Academy (Chelyabinsk)
* A total of three scheduled visits are planned during the course of this study. Visit 1 will occur during the Screening Period (Part A). Patients who enter the Screening Period (Part A) will be signing the ICF, instructed to follow regional dietary guidelines for the duration of the study. They will undergo clinical (biochemical, ultra-sound, duplex scan) and exercise SPECT imaging if applicable. Those individuals refusing to participate in the study will be taken into account with fixing the reason of unwillingness to participate.

All included subjects will be provided with a screening questionnaire querying the patient demographics, past medical history, patient FH history and diagnosis with FH type heterozygous or homozygous, family history of hypercholesterolemia, physical examination findings, current lipid-lowering therapies, and patients' contact information for further follow-up. After initialization of online data capture form (Electronic Medical System), the information will be also entered in the system.

For the patients with FH diagnosed on the basis of Dutch Lipid Clinic Network and/or Simon Broome Criteria or genetic testing Visit 2 will occur in a one month period. Visit 3 will occur in RussianCRPC in a one year±10 days period. At the scheduled visits update of the medical information, including monitoring of adverse cardiovascular events occurrence, changes in medications, and blood sampling, will be performed.

* Examination procedures at the scheduled visits:

  1. Signing the informed consent form (ICF)
  2. Filling the questionnaires to determine the classical cardiovascular risk factors, past medical history and treatment
  3. Applying Dutch Lipid Clinic Network (DLCN) and Simon Broome Register (SBR) criteria
  4. Maintaining Electronic Medical System by physicians participating in the Program
  5. Blood sampling for TC, triglycerides (TG), LDL-C, HDL-C, Lp(a), high-sensitivity C-reactive protein (hsCRP), PCSK9 measurement
  6. Genetic testing (mutations in the LDLR, apolipoprotein B (apoB), PCSK9 genes)
  7. Echocardiography for the assessment of ascending aorta and aortic valve
  8. Duplex scanning of the carotid arteries for the assessment of intima-media thickness and plaques' characteristics
  9. Exercise SPECT imaging in patients suspicious for coronary disease
  10. Annual evaluation of cardiovascular events (myocardial infarction, stroke, cardiovascular death, non-cardiovascular death, hospitalization due to acute coronary syndrome, heart failure, arterial revascularization procedures (percutaneous coronary intervention, coronary artery bypass grafting, endovascular or surgical revascularization in carotid arteries or lower extremities), aortic valve replacement.
* FH patients at these 1-st line Sites who meet inclusion criteria as described in the Methods section will be eligible to enroll. The same algorithm as described above will be initiated. Specialized staff from the Russian Cardiology Research and Production Complex (as a Core Center) will monitor the effectiveness and credibility of the undertaken work. Filling in the Electronic Medical System (eCRF) will be checked by the staff from the Core Center, and each year teleconferences will be held between the Sites-Participants of the Program.
* Perspectives: since 2018 ¬ the next phases of the Program will include recruitment of new set of Clinics, Policlinics and Institutions across Russia with specialized lipid clinics that could demonstrate acceptable feasibility for patient enrollment and engagement.

ELIGIBILITY:
Inclusion Criteria:

* Total cholesterol ≥7.5 mmol/L or LDL-C ≥4.9 mmol/L (pretreatment levels)
* Familial hypercholesterolemia defined as: a. Mutation in the LDL receptor and/or the ApoB gene and/or the PCSK9 gene; or b. clinical diagnosis of heterozygous FH (HeFH) according to the Dutch Lipid Network Criteria or Simon Broom Criteria
* Patients with genetic mutation of FH

Exclusion Criteria:

* uncontrolled primary hypothyroidism (thyroid stimulating hormone (TSH) >1.5 x upper limit of normal (ULN)),
* nephrotic syndrome and/or renal dysfunction (scrum creatinine >2.0 mg/dL or 160mmol/l, creatinine clearance <15 ml/min) at screening.
* uncontrolled diabetes mellitus (Glycated hemoglobin >8.5%)

Ages: 7 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Russian cohort of individuals who have been tested in the offices of the "INVITRO" Laboratory on the basis of advertising campaign for the purpose of total cholesterol level measurement and determination of cardiovascular risk with the use of SCORE chart.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2014-01; Primary Completion 2017-12-31 (Actual); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Prevalence of FH patients in the Russian Federation | at baseline

SECONDARY OUTCOMES:
Number of patients with heterozygous and homozygous forms of FH in Russia | at baseline
Distribution of lipoprotein(a) in individuals diagnosed with definite and probable FH. | at baseline
Severity of carotid atherosclerosis, aortic valve stenosis and coronary heart disease in Russian patients with FH | at baseline
  Assessment of carotid atherosclerosis will be performed with the use of carotid duplex scanning.
  Presence and severity of aortic valve stenosis will be evaluated with echocardiography.
  Exercise radionuclide myocardial perfusion imaging with single-photon emission computed tomography (SPECT) will be used for the diagnosis of myocardial ischemia in patients suspicious for CHD.
Mutations in following genes: low-density lipoprotein receptor (LDLR), proprotein convertase subtilisin/kexin type 9 (PCSK9), apolipoprotein B (apoB) | At baseline
  Genetic testing for FH-causing mutation in patients with probable and definite FH
Russian Registry of individuals with FH | up to 10 years
  Contribution in the formation of the Russian Health Ministry legislative acts concerning significance of FH as a socially and medically important disease with appropriate management strategies.
Prognosis of individuals with FH | at 1, 3, 5, 10 years
  Incidence of death from cardiovascular causes, nonfatal myocardial infarction, nonfatal stroke, revascularization procedures (cardiac, carotid, or peripheral), hospitalizations due to unstable angina pectoris or heart failure, all-cause mortality, diabetes in participants without baseline diabetes, new or recurrent cancers.

OTHER OUTCOMES:
Clinical and diagnostic significance of Dutch Lipid Clinic Network criteria and Simon Broome Registry criteria for diagnosis of FH in Russian population | up to 5 years
  Clinical and diagnostic significance of Dutch Lipid Clinic Network criteria and Simon Broome Registry criteria for the diagnosis of FH in Russia.
Family Health Team model and cascade testing in individuals with FH | up to 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Valery Kukharchuk, MD, DMSc, Study Chair — Russian Cardiology Research and Production Center; Igor Sergienko, MD, DMSc, Study Director — Russian Cardiology Research and Production Center; Marat Ezhov, MD, DMSc, Principal Investigator — Russian Cardiology Research and Production Center
Locations (5):
- Russia (5):
  - Chelyabinsk State Medical Academy, Chelyabinsk
  - EI Chazov National Medical Research Center of Cardiology, Moscow
  - Novosibirsk Research Institute of Internal Medicine, Institute of Internal Medicine Siberian Branch of the Russian Academy of Medical Sciences, Novosibirsk
  - Saint-Petersburg State University and North-West State Medical University n.a. I.I.Mechnikov, Saint Petersburg
  - Samara State Medical University, Samara

REFERENCES:
- [Background] M. S. Safarova, I. V. Sergienko, M. V. Ezhov, A. E. Semenova, M. A. Kachkovskiy, I. I. Shaposhnik, V. S. Gurevich, M. I. Voevoda, Y. P. Nikitin, V. V. Kuharchuk, Yu. A. Karpov Russian research program for early diagnosis and treatment of familial hypercholesterolaemia: Rationale and Design of the Russian FH Registry (RuFH). Journal of ATHEROSCLEROSIS AND DYSLIPIDAEMIAS 3: 7-15, 2014 (in Russian)
- [Background] Ezhov MV SI, Duplyakov DV, Abashina OE, Kachkovsky MA, Shaposhnik II, Genkel VV, Gurevich VS, Urazgildeeva SA, Tregubov AV, Konovalova TB, Muzalevskaya MV, Voevoda MI, Bazhan SS, Makarenkova KV, Timoshenko OV, Ragino YI, Urvantseva IA, Cozhocar KG, Sokolov AA, Boeva OI, Bolotova EV, Kushnaryova YB, Kuznetsova TY, Korneva VA, Bogdanov DY, Chichina EE, Soloviev VM, Smolenskaya OG, Galyavich AS, Safarova MS, Popova AV, Malakhov VV, Ansheles AA, Nozadze DN, Semenova AE, Rozhkova TA, Solovéva EY, Gornyakova NB, Karpov YA, Kukharchuk VV. Results of the Russian research program on the diagnosis and treatment of patients with familial hypercholesterolemia. High prevalence, low awareness, poor adherence. Atherosclerosis and Dyslipidaemias An official Journal of the Russian National Atherosclerosis Society (RNAS) 2017;2:5-15.
- [Result] EAS Familial Hypercholesterolaemia Studies Collaboration, Vallejo-Vaz AJ, Akram A, Kondapally Seshasai SR, Cole D, Watts GF, Hovingh GK, Kastelein JJ, Mata P, Raal FJ, Santos RD, Soran H, Freiberger T, Abifadel M, Aguilar-Salinas CA, Alnouri F, Alonso R, Al-Rasadi K, Banach M, Bogsrud MP, Bourbon M, Bruckert E, Car J, Ceska R, Corral P, Descamps O, Dieplinger H, Do CT, Durst R, Ezhov MV, Fras Z, Gaita D, Gaspar IM, Genest J, Harada-Shiba M, Jiang L, Kayikcioglu M, Lam CS, Latkovskis G, Laufs U, Liberopoulos E, Lin J, Lin N, Maher V, Majano N, Marais AD, März W, Mirrakhimov E, Miserez AR, Mitchenko O, Nawawi H, Nilsson L, Nordestgaard BG, Paragh G, Petrulioniene Z, Pojskic B, Reiner Ž, Sahebkar A, Santos LE, Schunkert H, Shehab A, Slimane MN, Stoll M, Su TC, Susekov A, Tilney M, Tomlinson B, Tselepis AD, Vohnout B, Widén E, Yamashita S, Catapano AL, Ray KK. Pooling and expanding registries of familial hypercholesterolaemia to assess gaps in care and improve disease management and outcomes: Rationale and design of the global EAS Familial Hypercholesterolaemia Studies Collaboration. Atheroscler Suppl. 2016;22:1-32. doi: 10.1016/j.atherosclerosissup.2016.10.001.